CLINICAL TRIAL: NCT04184739
Title: Investigating the Quality and Effectiveness of a Personalised Mobile App Designed to Support Patients With Fixed (Train Track) Braces: A Randomised Controlled Trial (Student Study)
Brief Title: Quality and Effectiveness of a Personalised App to Support Patients With Fixed Braces
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 124581
Record Dates: First submitted 2019-11-19; First posted 2019-12-04 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-11

CONDITIONS: Treatment Adherence and Compliance
MeSH Terms: conditions — Treatment Adherence and Compliance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Active Comparator): Standard treatment information (verbal and written) and access to a basic version of the App with a toothbrushing timer. The timer is necessary as the health behaviour outcome is toothbrushing duration.
  Interventions: Other: My Braces App
- Group B (Experimental): As for group A, however, additionally the App will provide generic treatment information (a combination of videos and text)
  Interventions: Other: My Braces App
- Group C (Experimental): As for group B, however, the patients will have access to the full functionality of the App and the App will allow patients to input their own personalised treatment information (including progress photographs), set goals, develop plans for achieving these and provide the patient and clinicians with appropriate dashboards to monitor progress.
  Interventions: Other: My Braces App

INTERVENTIONS:
Other: My Braces App — An App designed to support patients undertaking orthodontic treatment.

SUMMARY:
Mobile phones are potentially an invaluable tool in improving adherence, they are readily available and can utilised to deliver several approaches to improve adherence simultaneously. A personalised App to help support orthodontic patients ('My Braces') was therefore developed by the researchers. The App provides generic treatment information and also has a personalised element. The personalised element allows patients to input their own treatment information (including progress photographs), set goals, develop plans for achieving these and it provides the patient and clinicians with appropriate dashboards to monitor progress.

This research will be conducted at the Eastman Dental Hospital, UCLH Foundation Trust, London. The aim is to assess the effectiveness of the My Braces App, an App designed to support patients undergoing fixed orthodontic treatment.

Effectiveness of the My Braces App will be tested by way of a randomised controlled trial. Participants will be allocated to one of three groups:

Group A: Standard treatment information (verbal and written) and access to a basic version of the My Braces App with a toothbrushing timer. The timer is necessary as the health behaviour outcome is toothbrushing duration.

Group B: As for group A, however, additionally the My Braces App will provide generic treatment information (a combination of videos and text)

Group C: As for group B, however, the patients will have access to the full functionality of the My Braces App and the App will allow patients to input their own personalised treatment information (including progress photographs), set goals, develop plans for achieving these and provide the patient and clinicians with appropriate dashboards to monitor progress.

DETAILED DESCRIPTION:
The National Child Dental Health Survey (England, Wales and Northern Ireland) indicated that 9% of 12 years olds are receiving orthodontic treatment (the use of braces to straighten teeth) and a further 37% have an unmet need. Treatment duration is lengthy (2-3 years on average) and adherence to treatment advice is essential for successful outcomes. It has been reported that up to 43% of patients fail to complete treatment and there are currently no useful predictors of non-completion. The NHS England annual spend on primary care orthodontics is in excess of £200 million, non-completion of treatment therefore represents a significant inefficient use of public resources.

Mobile phones are potentially an invaluable tool in improving adherence, they are readily available and can utilised to deliver several approaches to improve adherence simultaneously. A personalised App to help support orthodontic patients ('My Braces') was therefore developed by the researchers. The App provides generic treatment information and also has a personalised element. The personalised element allows patients to input their own treatment information (including progress photographs), set goals, develop plans for achieving these and it provides the patient and clinicians with appropriate dashboards to monitor progress.

This research will be conducted at the Eastman Dental Hospital, UCLH Foundation Trust, London. The aim is to assess the effectiveness of the My Braces App, an App designed to support patients undergoing fixed orthodontic treatment.

Effectiveness of the My Braces App will be tested by way of a randomised controlled trial. Participants will be allocated to one of three groups:

Group A: Standard treatment information (verbal and written) and access to a basic version of the My Braces App with a toothbrushing timer. The timer is necessary as the health behaviour outcome is toothbrushing duration.

Group B: As for group A, however, additionally the My Braces App will provide generic treatment information (a combination of videos and text)

Group C: As for group B, however, the patients will have access to the full functionality of the My Braces App and the App will allow patients to input their own personalised treatment information (including progress photographs), set goals, develop plans for achieving these and provide the patient and clinicians with appropriate dashboards to monitor progress.

It is important to include Group B as this will allow the team to ascertain whether it is the personalisation of the App content which infers any benefit over and above providing generic information via an App if a difference is found between Groups A and C.

ELIGIBILITY:
Inclusion Criteria:

* Patients accepted for orthodontic treatment utilising fixed orthodontic braces ('train track' braces) at the Eastman Dental Hospital, UCLH Foundation Trust (UCLH EDH)
* 10-18 years (inclusive) at the start of treatment
* Familiarity with, and daily access to, a smartphone/tablet • Ability to read and communicate in English

Exclusion Criteria:

* Craniofacial/Orthognathic patients or those with severe hypodontia (developmental absence of teeth); these patients require complex multi-disciplinary treatment. The information need for these patients is therefore different to routine orthodontic treatment
* Communication difficulties (for example, severe autism, learning difficulties)
* Patients who are aware that a family member/friend is enrolled in the study (including a preceding feasibility study, the pilot or RCT) - this is to avoid the patient potentially having access to parts of the App relating to groups other than that the patient is allocated to

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 138 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Toothbrushing duration | 3 months
  Timed toothbrush use will be determined via the information stored on the App. It is anticipated that participants will not remember to time each brushing episode, therefore, the duration and number of brushing sessions stored within the App will allow for the average brushing duration to be determined. The unit of measurement will be seconds.
Toothbrushing duration | 12 months
  Timed toothbrush use will be determined via the information stored on the App. It is anticipated that participants will not remember to time each brushing episode, therefore, the duration and number of brushing sessions stored within the App will allow for the average brushing duration to be determined. The unit of measurement will be seconds.
Toothbrushing duration | End of treatment (24-36 months on average)
  Timed toothbrush use will be determined via the information stored on the App. It is anticipated that participants will not remember to time each brushing episode, therefore, the duration and number of brushing sessions stored within the App will allow for the average brushing duration to be determined. The unit of measurement will be seconds.
Bleeding score | Base line (start of treatment)
  A periodontal probe will be utilised, the presence of bleeding within 10 to 30 seconds of probing is indicative of inflammation of the gingivae. Scores will be recorded for all teeth anterior to the molars (incisors, canines and premolars) and will be recorded as the percentage of the total number of tooth surfaces (6 aspects per tooth). A binary score will be assigned to each surface (1 bleeding present, 0 no bleeding).
Bleeding score | 3 months
  A periodontal probe will be utilised, the presence of bleeding within 10 to 30 seconds of probing is indicative of inflammation of the gingivae. Scores will be recorded for all teeth anterior to the molars (incisors, canines and premolars) and will be recorded as the percentage of the total number of tooth surfaces (6 aspects per tooth). A binary score will be assigned to each surface (1 bleeding present, 0 no bleeding).
Bleeding score | 12 months
  A periodontal probe will be utilised, the presence of bleeding within 10 to 30 seconds of probing is indicative of inflammation of the gingivae. Scores will be recorded for all teeth anterior to the molars (incisors, canines and premolars) and will be recorded as the percentage of the total number of tooth surfaces (6 aspects per tooth). A binary score will be assigned to each surface (1 bleeding present, 0 no bleeding).
Bleeding score | End of treatment (24-36 months on average)
  A periodontal probe will be utilised, the presence of bleeding within 10 to 30 seconds of probing is indicative of inflammation of the gingivae. Scores will be recorded for all teeth anterior to the molars (incisors, canines and premolars) and will be recorded as the percentage of the total number of tooth surfaces (6 aspects per tooth). A binary score will be assigned to each surface (1 bleeding present, 0 no bleeding).

SECONDARY OUTCOMES:
Plaque score | Base line (start of treatment), 3 months, 12 months, and at the end of treatment (24-36 months on average)
  Plaque scores will be recorded for all teeth anterior to the molars (incisors, canines and premolars) as the percentage of total surfaces (6 aspects per tooth). A plaque disclosing agent will be used for the plaque assessment. A binary score will be assigned to each surface (1 plaque present, 0 no plaque present).
Number of breakages | 3 months, 12 months, and at the end of treatment (24-36 months on average)
  Information relating to the number of breakages will be obtained from the patient's medical records.
Number of missed appointments | 3 months, 12 months, and at the end of treatment (24-36 months on average)
  Information relating to the number of missed appointments will be obtained from the patient's medical records.
Total number of appointments | At the end of treatment (24-36 months on average)
  Information relating to the number of missed or rescheduled appointments and emergency appointments will be obtained from the patient's medical records.
Treatment duration | At the end of treatment (24-36 months on average)
  Information relating to treatment duration will be obtained from the patient's medical records.
Enamel demineralisation on the front 6 teeth using standardised photographs | Base line (start of treatment) and at the end of treatment (24-36 months on average)
  For the evaluation of demineralisation, photographs will be assessed and the severity of enamel demineralization will be recorded. The labial surfaces of the upper incisors and canines will be scored as follows:
  1. No white spot formation
  2. Slight white spot formation (thin rim)
  3. Excessive white spot formation (thicker bands) 4. White spot formation with cavitation
App subjective quality | 3 months and at the end of treatment (24-36 months on average)
  Patients will be asked to complete sections E and F of the uMARS questionnaire to ascertain perceived App quality.
App engagement (pages accessed and whether this changes with time) | 3 months, 12 months, and at the end of treatment (24-36 months on average)
  Data relating to App usage will be obtained from the Google Firebase system.

CONTACTS AND LOCATIONS:
Overall Officials: Susan J Cunningham, PhD, Principal Investigator — UCL Professor

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sharif MO, Newton JT, Cunningham SJ. Assessing the Effectiveness and Acceptability of a Personalized Mobile Phone App in Improving Adherence to Oral Hygiene Advice in Orthodontic Patients: Protocol for a Feasibility Study and a Randomized Controlled Trial. JMIR Res Protoc. 2021 Jan 13;10(1):e18021. doi: 10.2196/18021. PMID 33439142